CLINICAL TRIAL: NCT00166309
Title: FENOC: The FEIBA NovoSeven Comparative Study
Brief Title: The FEIBA NovoSeven Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FENOC
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Severe Hemophilia A With an Inhibitor
Keywords: Hemophilia A; Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — anti-inhibitor coagulant complex; recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: FEIBA and NovoSeven

SUMMARY:
FENOC is a prospective, open-label, randomized, cross-over, multi-center study to investigate and compare the hemostatic effect and cost-efficacy of two different by-passing agents in the treatment of joint hemorrhages in subjects with severe hemophilia A and inhibitors. The study is designed as a clinical equivalency trial.

DETAILED DESCRIPTION:
The incidence of inhibitors among people with severe hemophilia A has been documented as approximately 20-30% in several prospective studies. In such patients acute hemorrhages frequently occur and profoundly jeopardize health, with subsequent development of arthropathy. A common way of treating such bleeding episodes is to use bypassing agents. Among these agents the prothrombin complex concentrate FEIBA has been widely used for many years. More recently, recombinant factor VIIa (NovoSeven) has been added to the therapeutic options. While both products have been found effective in treating hemorrhages, the number of injections given for a bleeding episode has ranged widely, and it is so far unknown whether one of the products might have a better effect in certain patients.

ELIGIBILITY:
Inclusion Criteria:

* Congenital hemophilia A with an inhibitor and the need for by-passing agents in the case of joint bleeding.
* An expected bleeding frequency of >=3 joint bleeds per year.
* Informed consent given.
* Age of two or older.

Exclusion Criteria:

* Other congenital and acquired bleeding disorders.
* Symptomatic liver disease.
* Life expectancy <12 months.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2000-07; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
-The hemostatic effect of treatment with a single dose of FEIBA with that of two doses of NovoSeven on joint hemorrhages after 6 hours.

SECONDARY OUTCOMES:
The hemostatic effect of treatment after 2, 12, 24 36, and 48 hours.
The difference in pain, rated using the 100 mm visual analog scale (VAS) before treatment and after 2 (before the second dose of NovoSeven, 6, 12, 24, 36, and 48 hours.
The number of infusions required of each concentrate to stop the bleeding.
The use of analgesics.
Cost-efficacy, analyzed on the basis of clinical response.
Correlation between thrombin generation in vitro with each concentrate and the in vivo clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Berntorp, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Malmo University Hospital, Malmo, Sweden

REFERENCES:
- [Result] Astermark J, Donfield SM, DiMichele DM, Gringeri A, Gilbert SA, Waters J, Berntorp E; FENOC Study Group. A randomized comparison of bypassing agents in hemophilia complicated by an inhibitor: the FEIBA NovoSeven Comparative (FENOC) Study. Blood. 2007 Jan 15;109(2):546-51. doi: 10.1182/blood-2006-04-017988. Epub 2006 Sep 21. PMID 16990605